CLINICAL TRIAL: NCT02442856
Title: Non-invasive Measurement of Cerebral Dynamic Autoregulation
Acronym: TOMCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 821705
Record Dates: First submitted 2015-05-08; First posted 2015-05-13 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): We will measure dCA with both TCD and DCS during acute changes in mean arterial pressure using thigh cuff deflation techniques in vascular risk factor subjects. Measurements will be compared between TCD and DCS in order to validate DCS as a tool to measure dCA in this population.
  Interventions: Device: Thigh Cuff

INTERVENTIONS:
Device: Thigh Cuff

SUMMARY:
The overall objective of this study is to evaluate the use of diffuse correlation spectroscopy to non-invasively measure dynamic cerebral autoregulation in subjects with vascular risk factors. Optical cerebral blood flow measurements will be correlated with changes in arterial blood pressure to assess how CBF is maintained in response to changes in ABP, and will be compared to transcranial doppler reference measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 50 years
* Positive history of at least one of the following vascular disk factors: hypertension, diabetes, hyperlipidemia, coronary artery disease, atrial fibrillation, prior myocardial infarct, transient ischemic attack, or history of smoking

Exclusion Criteria:

* Vascular risk factor subjects:

  1. Pregnant women
  2. Prisoners
  3. Prior neurosurgical procedure or traumatic brain injury, including hemicraniectomy or other skull defect
  4. Prior history of ischemic or hemorrhagic stroke
  5. Prior lower extremity amputation
  6. Peripheral vascular disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: We will measure dynamic cerebral autoregulation (dCA) with both transcranial doppler (TCD) and diffuse correlation spectroscopy (DCS) during acute changes in mean arterial pressure using thigh cuff deflation techniques in vascular risk factor subjects. Measurements will be compared between TCD and DCS in order to validate DCS as a tool to measure dCA in this population.
Period: Overall Study
Arm/Group | Intervention
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 21
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 31 [29 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: dCA Measurement During Acute Changes in Mean Arterial Pressure, TCD
Description: Rate of Regulation, measured using transcranial doppler. Rate of regulation (ROR) is calculated as follows: ROR = (change in relative cerebrovascular resistance / change in time) / maximum fractional decrease in blood pressure due to thigh cuff deflation.
Time Frame: 1.5 hours
Population: 21 subjects consented, hemodynamic monitoring possible in 18. 1 subject did not tolerate,data acquisition was unsuccessful in 2. In 3 subjects, the pressure algorithm to isolate cerebral blood flow(CBF) was unsuccessful. In 4 subjects, BP did not decrease following cuff deflation due to technical issues leaving 11 subjects in the final analysis
Measure: Number (95% Confidence Interval); unit: per second
Arm/Group | Intervention
Number analyzed (Participants) | 11
per second | 0.262 [0.170 to 0.366]

2. Primary Outcome: dCA Measurement During Acute Changes in Mean Arterial Pressure, Optical
Description: Rate of Regulation, measured using diffuse correlation spectroscopy. Rate of regulation (ROR) is calculated as follows: ROR = (change in relative cerebrovascular resistance / change in time) / maximum fractional decrease in blood pressure due to thigh cuff deflation.
Time Frame: 1.5 hours
Population: 21 subjects in the study, but hemodynamic monitoring was only possible in 18. 1 subject did not tolerate, and data acquisition was unsuccessful in 2. In 3 subjects, the pressure algorithm to isolate CBF was unsuccessful. In 4 subjects, BP did not decrease following cuff deflation due to technical issues leaving 11 subjects in the final analysis
Measure: Number (95% Confidence Interval); unit: per second
Arm/Group | Intervention
Number analyzed (Participants) | 11
per second | 0.278 [0.199 to 0.300]

3. Other Pre Specified Outcome: Linear Relationship Between Rate of Regulation Measured Using TCD and Optics
Description: Linear relationship between Rate of Regulation measured using TCD and Optics, expressed as slope of linear fit
Time Frame: 1.5 hours
Measure: Number; unit: slope
Arm/Group | Intervention
Number analyzed (Participants) | 11
slope | 0.96

ADVERSE EVENTS:
Time Frame: Duration of study, which was approximately 6 months.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-03-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT02442856/Prot_SAP_ICF_000.pdf